CLINICAL TRIAL: NCT00010803
Title: Ginkgo Biloba Prevention Trial in Older Individuals
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: Office of Dietary Supplements (ODS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute on Aging (NIA) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: U01 AT000162-01M; U01AT000162-01 (NIH); NCT00004535 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Results first posted 2010-09-16 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Dementia; Alzheimer's Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — Ginkgo Extract; Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo 1 pill twice a day
  Interventions: Drug: Placebo
- Ginkgo biloba (Active Comparator): Ginkgo biloba EGb761 120 mg twice daily
  Interventions: Drug: Ginkgo biloba

INTERVENTIONS:
Drug: Ginkgo biloba — 120mg twice a day
  Other Names: EGb761
  Arms: Ginkgo biloba
Drug: Placebo — One pill twice daily
  Other Names: Identical appearance as Ginkgo biloba pill
  Arms: Placebo

SUMMARY:
This study will determine the effect of 240mg/day Ginkgo biloba in decreasing the incidence of dementia and specifically Alzheimer's disease (AD), slowing cognitive decline and functional disability, reducing incidence of cardiovascular disease, and decreasing total mortality.

DETAILED DESCRIPTION:
Participants will be studied in a randomized trial of 240 mg of Ginkgo biloba as compared to placebo in healthy men and women, at least 75 years old. The trial will last approximately 8 years. The intervention will be considered unsuccessful in those participants who succumb to dementia, including Alzheimer's Disease and vascular dementia. There are four clinical centers: Pittsburgh, PA; Hagerstown, MD; Winston-Salem, NC; and Sacramento, CA; and a Coordinating Center at the University of Washington, Seattle. There will be a clinic visit every 6 months to determine morbidity, mortality and change in cognition that will include repeat of ADAS, CDR, and 10 battery neuropsychological evaluation and informant interview. The primary endpoint is dementia, specifically Alzheimer's disease, secondary endpoint will include the incidence of vascular disease, changes in cognitive function scores over time, total mortality and changes in functional status. The diagnosis of dementia will be based on neuropsychological testing, neurological exam, MRI, functional measurements, and review by a central adjudication committee and classified by DSM IV, NINCDS criteria and ADRTC criteria for vascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Non-demented participants
* Willing to participate in a seven-year follow-up trial of Ginkgo Biloba
* English is their usual language
* Willing informant who has frequent contact with the participant

Exclusion Criteria:

* Currently on anticoagulant therapy
* Cancer diagnosed and treated within the past two years (except for skin cancer)
* Participant with class III - IV congestive heart failure
* Currently being treated with psychopharmacological drugs for depression
* Hospitalized for depression within the last year
* Taking Aricept (or similar agents) for cognitive problems or dementia
* Baseline blood creatinine >2
* Baseline SGGT is a marker of liver function (3 x normal>or=90 IU)
* Baseline hematocrit<30
* Baseline white blood count>or=15,000

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 3069 (Actual)
Dates: Start 2000-10; Primary Completion 2008-04 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven T. DeKosky, M.D., Principal Investigator — University of Pittsburgh, Department of Neurology
Locations (5):
- United States (5):
  - University of California, Davis, Sacramento, California
  - Johns Hopkins University, Baltimore, Maryland
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Pittsburgh/University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Background] Fitzpatrick AL, Fried LP, Williamson J, Crowley P, Posey D, Kwong L, Bonk J, Moyer R, Chabot J, Kidoguchi L, Furberg CD, DeKosky ST; GEM Study Investigators. Recruitment of the elderly into a pharmacologic prevention trial: the Ginkgo Evaluation of Memory Study experience. Contemp Clin Trials. 2006 Dec;27(6):541-53. doi: 10.1016/j.cct.2006.06.007. Epub 2006 Jul 4. PMID 16949348
- [Background] DeKosky ST, Fitzpatrick A, Ives DG, Saxton J, Williamson J, Lopez OL, Burke G, Fried L, Kuller LH, Robbins J, Tracy R, Woolard N, Dunn L, Kronmal R, Nahin R, Furberg C; GEMS Investigators. The Ginkgo Evaluation of Memory (GEM) study: design and baseline data of a randomized trial of Ginkgo biloba extract in prevention of dementia. Contemp Clin Trials. 2006 Jun;27(3):238-53. doi: 10.1016/j.cct.2006.02.007. Epub 2006 Apr 19. PMID 16627007
- [Background] Fitzpatrick AL, Buchanan CK, Nahin RL, Dekosky ST, Atkinson HH, Carlson MC, Williamson JD; Ginkgo Evaluation of Memory (GEM) Study Investigators. Associations of gait speed and other measures of physical function with cognition in a healthy cohort of elderly persons. J Gerontol A Biol Sci Med Sci. 2007 Nov;62(11):1244-51. doi: 10.1093/gerona/62.11.1244. PMID 18000144
- [Background] Nahin RL, Fitzpatrick AL, Williamson JD, Burke GL, Dekosky ST, Furberg C; GEM Study Investigators. Use of herbal medicine and other dietary supplements in community-dwelling older people: Baseline data from the ginkgo evaluation of memory study. J Am Geriatr Soc. 2006 Nov;54(11):1725-35. doi: 10.1111/j.1532-5415.2006.00942.x. PMID 17087700
- [Background] Rosano C, Aizenstein HJ, Cochran JL, Saxton JA, De Kosky ST, Newman AB, Kuller LH, Lopez OL, Carter CS. Event-related functional magnetic resonance imaging investigation of executive control in very old individuals with mild cognitive impairment. Biol Psychiatry. 2005 Apr 1;57(7):761-7. doi: 10.1016/j.biopsych.2004.12.031. PMID 15820233
- [Background] Rosano C, Aizenstein H, Cochran J, Saxton J, De Kosky S, Newman AB, Kuller LH, Lopez OL, Carter CS. Functional neuroimaging indicators of successful executive control in the oldest old. Neuroimage. 2005 Dec;28(4):881-9. doi: 10.1016/j.neuroimage.2005.05.059. Epub 2005 Oct 12. PMID 16226041
- [Background] Williamson JD, Vellas B, Furberg C, Nahin R, Dekosky ST. Comparison of the design differences between the Ginkgo Evaluation of Memory study and the GuidAge study. J Nutr Health Aging. 2008 Jan;12(1):73S-9S. doi: 10.1007/BF02982591. PMID 18165850
- [Background] Saxton J, Snitz BE, Lopez OL, Ives DG, Dunn LO, Fitzpatrick A, Carlson MC, Dekosky ST; GEM Study Investigators. Functional and cognitive criteria produce different rates of mild cognitive impairment and conversion to dementia. J Neurol Neurosurg Psychiatry. 2009 Jul;80(7):737-43. doi: 10.1136/jnnp.2008.160705. Epub 2009 Mar 11. PMID 19279031
- [Background] Snitz BE, Saxton J, Lopez OL, Ives DG, Dunn LO, Rapp SR, Carlson MC, Fitzpatrick AL, Dekosky ST; GEM study Investigators. Identifying mild cognitive impairment at baseline in the Ginkgo Evaluation of Memory (GEM) study. Aging Ment Health. 2009 Mar;13(2):171-82. doi: 10.1080/13607860802380656. PMID 19347684
- [Result] DeKosky ST, Williamson JD, Fitzpatrick AL, Kronmal RA, Ives DG, Saxton JA, Lopez OL, Burke G, Carlson MC, Fried LP, Kuller LH, Robbins JA, Tracy RP, Woolard NF, Dunn L, Snitz BE, Nahin RL, Furberg CD; Ginkgo Evaluation of Memory (GEM) Study Investigators. Ginkgo biloba for prevention of dementia: a randomized controlled trial. JAMA. 2008 Nov 19;300(19):2253-62. doi: 10.1001/jama.2008.683. PMID 19017911
- [Result] Kuller LH, Ives DG, Fitzpatrick AL, Carlson MC, Mercado C, Lopez OL, Burke GL, Furberg CD, DeKosky ST; Ginkgo Evaluation of Memory Study Investigators. Does Ginkgo biloba reduce the risk of cardiovascular events? Circ Cardiovasc Qual Outcomes. 2010 Jan;3(1):41-7. doi: 10.1161/CIRCOUTCOMES.109.871640. Epub 2009 Nov 24. PMID 20123670
- [Result] Snitz BE, O'Meara ES, Carlson MC, Arnold A, Ives DG, Rapp SR, Saxton J, Lopez OL, Dunn LO, Sink K, DeKosky ST for the Ginkgo Evaluation of Memory Study investigators. Ginkgo biloba in preventing cognitive decline in older adults: A randomized trial. Journal of the American Medical Aassociation, 2009, in press.
- [Derived] Snitz BE, O'Meara ES, Carlson MC, Arnold AM, Ives DG, Rapp SR, Saxton J, Lopez OL, Dunn LO, Sink KM, DeKosky ST; Ginkgo Evaluation of Memory (GEM) Study Investigators. Ginkgo biloba for preventing cognitive decline in older adults: a randomized trial. JAMA. 2009 Dec 23;302(24):2663-70. doi: 10.1001/jama.2009.1913. PMID 20040554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occured between September 2000 through June 2002 primarily using mass mailings from targeted lists such as voter's registration and commercially available lists. Some sites chose to supplement this approach with newspaper, radio and television ads plus newsletter articles, posters and community presentations.
Pre-assignment Details: After mailing brochures to potential participants, we conducted a telephone screening followed by an in-person clinic visit to finalize eligibility. Randomization was done at a second visit within close proximity to the screening visit.
Groups:
- Ginkgo Biloba: EGb 761 Ginkgo biloba 120 mg twice daily
- Placebo: Placebo twice daily
Period: Overall Study
Arm/Group | Ginkgo Biloba | Placebo
Started | 1545 (Randomized) | 1524 (Randomized)
Completed | 1448 (Reached endpoint of dementia, death or completion) | 1426 (Reached endpoint of dementia, death or completion)
Not Completed | 97 | 98
Not completed — Withdrawal by Subject | 97 | 98

BASELINE CHARACTERISTICS:
Groups:
- Ginkgo Biloba: 120 mg twice daily, total 240 mg
- Placebo: Placebo 1 pill twice daily
- Total: Total of all reporting groups
Arm/Group | Ginkgo Biloba | Placebo | Total
Number analyzed (Participants) | 1545 | 1524 | 3069
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1545 | 1524 | 3069
Age Continuous [Mean (Standard Deviation); unit: years] | 79.1 (3.3) | 79.1 (3.3) | 79.1 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 702 | 716 | 1418
  Male | 843 | 808 | 1651
Region of Enrollment [Number; unit: participants]
  United States | 1545 | 1524 | 3069

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incident Dementia
Description: All cause dementia based on DSM-IV criteria as determined by an expert panel of clinicians using an adjudication process. A full neuropsychological battery was administered annually, or at 6 month visit if there was a diagnosis of dementia or initiation of medication for dementia by private physician, or change in Modified Mini Mental State Exam (3MSE), Clinical Dementia Rating (CDR), or Alzheimer Disease Assessment Scale (ADAS-Cog). Decline on tests scores based on an algorithm resulted in a neurological exam and brain imaging. These data were used in the adjudication process.
Time Frame: Brief neuropsychological testing every 6 months, detailed testing annually, average 6.1 years follow up
Population: Subjects developing incident dementia during trial in each group, intention to treat (ITT).
Measure: Number; unit: Participants
Arm/Group | Ginkgo Biloba | Placebo
Number analyzed (Participants) | 1545 | 1524
Participants | 277 | 246
Statistical Analysis 1: Comparison: Ginkgo Biloba vs Placebo; The null hypothesis is that the instantaneous hazard rate for Ginkgo biloba and placebo are the same. Assumptions were based on 4%/yr dementia and 6%/yr mortality and dropout combined. A sample size of 3000 with an average follow up of 5 years resulted in 96% power to detecting a 30% reduction in the rate of dementia at a 2-sided significance level of 0.5; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.21, Log Rank; Time to dementia in Ginkgo vs placebo groups. The Cox proportional hazards model was used to compute hazard ratios and log-rank tests; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.94 to 1.33]

2. Secondary Outcome: Number of Participants With the Indicated Cardiovascular Disease or Mortality
Description: Myocardial infarction (MI), angina, stroke (CVA), transient ischemic attack (TIA), combined coronary heart disease (CHD) (MI/angina), combined cerebrovascular (CVA/TIA), peripheral vascular disease, and mortality
Time Frame: 6 months
Population: Total cohort of 3069 based on same design as primary outcome, ITT.
Measure: Number; unit: Participants
Arm/Group | Ginkgo Biloba | Placebo
Number analyzed (Participants) | 1545 | 1524
Participants
  Total Mortality | 197 | 188
  Atherosclerotic CHD Mortality | 45 | 42
  Incident MI | 68 | 60
  Incident Angina | 66 | 76
  Incident CHD (MI &/or angina) | 107 | 110
  Incident CHF | 112 | 122
  Incident Stroke | 73 | 59
  Incident TIA | 27 | 31
  Incident CVD (stroke &/or TIA) | 99 | 88
  Total CHD and CVD | 157 | 154
Statistical Analysis 1: Comparison: Ginkgo Biloba vs Placebo; Total Mortality; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.70, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.85 to 1.27]
Statistical Analysis 2: Comparison: Ginkgo Biloba vs Placebo; Atherosclerotic CHD mortality; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.78, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.70 to 1.62]
Statistical Analysis 3: Comparison: Ginkgo Biloba vs Placebo; Incident Myocardial Infarction; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.54, Log Rank; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.79 to 1.58]
Statistical Analysis 4: Comparison: Ginkgo Biloba vs Placebo; Incident Angina; Test type: Non-Inferiority or Equivalence — Previously Provided; p = 0.32, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.61 to 1.18]
Statistical Analysis 5: Comparison: Ginkgo Biloba vs Placebo; Incident CHD; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.66, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.72 to 1.23]
Statistical Analysis 6: Comparison: Ginkgo Biloba vs Placebo; Incident CHF; Test type: Non-Inferiority or Equivalence — Previously Provided; p = 0.48, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.71 to 1.18]
Statistical Analysis 7: Comparison: Ginkgo Biloba vs Placebo; Incident Stroke; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.25, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.52 to 1.45]
Statistical Analysis 8: Comparison: Ginkgo Biloba vs Placebo; Incident TIA; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.59, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.52 to 1.45]
Statistical Analysis 9: Comparison: Ginkgo Biloba vs Placebo; Incident CVD; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.42, Log Rank; Cox Proportional Hazard = 1.12, 95% CI 2-sided [0.84 to 1.50]
Statistical Analysis 10: Comparison: Ginkgo Biloba vs Placebo; Total CHD and CVD combined; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.98, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.80 to 1.25]

3. Secondary Outcome: Progression of Cognitive Decline in Standardized Z-score Scale. Higher Z-scores Indicate Worse Performance.
Description: Rate of annual change by cognitive domain in standardized Z-score scale. Higher Z-scores indicate worse performance. Best score = -2.0 Z-score change per year (improvement); worse score = 2.0 Z-score change per year (decline).
Time Frame: 6 months/annually
Population: Final test scores were imputed for participants who did not have a cognitive exam during the year before death (n=234) or dropout (n=154) or during the month before censoring for dementia (n=70). Factors in imputed model included treatment group, demographic and health history variables, study site, and other cognitive scores. Higher Z-scores worse
Measure: Mean (95% Confidence Interval); unit: Z-score units
Arm/Group | Ginkgo Biloba | Placebo
Number analyzed (Participants) | 1545 | 1524
Z-score units
  Global Cognition (mean Z-score of 5 domains) | 0.069 [0.064 to 0.074] | 0.071 [0.065 to 0.076]
  Memory (mean Z-score of 2 memory tests) | 0.043 [0.034 to 0.051] | 0.041 [0.032 to 0.050]
  Attention (mean Z-score of 2 attention tests) | 0.043 [0.037 to 0.050] | 0.048 [0.041 to 0.054]
  Visuospatial Abilities (mean Z-score of 2 tests) | 0.107 [0.097 to 0.117] | 0.118 [0.108 to 0.128]
  Language (mean Z-score of 2 language tests) | 0.045 [0.037 to 0.054] | 0.041 [0.033 to 0.048]
  Executive Functions (mean Z-score of 2 tests) | 0.092 [0.086 to 0.099] | 0.089 [0.082 to 0.096]
Statistical Analysis 1: Comparison: Ginkgo Biloba vs Placebo; Linear mixed models comparing rates of change in global cognition scores (z-scores) by treatment group; Test type: Superiority or Other; p = .65, Mixed Models Analysis; Treatment X Time interaction = -0.002, 95% CI 2-sided [-0.009 to 0.005]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected every six months at testing visits, and at interim 3 month adherence phone calls.
Arm/Group | Ginkgo Biloba | Placebo
Serious Adverse Events (participants affected / at risk) | 1000/1545 | 961/1524
Other Adverse Events (participants affected / at risk) | 1504/1545 | 1469/1524
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ginkgo Biloba (N=1545) | Placebo (N=1524)
Death (General disorders) | 197 (197) | 188 (188)
Bleeding (General disorders) | 138 (171) | 140 (178) — Gastrointestinal and all other
Coronary Heart Disease Total (Vascular disorders) | 211 (285) | 204 (259) — Myocardial infarction, angina, angioplasty, coronary artery bypass graft, coronary heart disease death
Stroke (Vascular disorders) | 80 (88) | 71 (82) — Ischemic, hemorrhagic and unknown
All other SAEs (General disorders) | 374 (1627) | 358 (1647)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ginkgo Biloba (N=1545) | Placebo (N=1524)
non-hospitalized self-reported symptom (General disorders) | 0 (0) | 0 (0)
All adverse events (General disorders) | 1504 (1504) | 1469 (1469) — There were no statistically significant differences.
Self-reported non-hospitalized symptom collected every 6 months (General disorders) | 1504 (1504) | 1469 (1469)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No